CLINICAL TRIAL: NCT02252029
Title: RotaNeo: Evaluation of Rotavirus Vaccine Administration in Premature Babies in the Neonatal Unit
Brief Title: Rotavirus Vaccine in Premature Babies
Acronym: RotaNeo
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: OVG 2014/04
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Gastroenteritis
Keywords: Rotavirus; Vaccine
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool, serum
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will establish the duration of excretion of rotavirus vaccine in stool following vaccination of premature babies hospitalised in a neonatal unit at the time of vaccination.

DETAILED DESCRIPTION:
Rotavirus is the commonest cause of severe gastroenteritis in young children, and premature babies are at high risk of serious disease. The RV1 rotavirus vaccine is an altered form of the virus and is given to all children at 8 weeks and 12 weeks of age in the UK. It is given by mouth and excreted in the stool following vaccination - the vaccine virus can therefore be transmitted between people in the same way as the normal virus. Premature babies often receive their initial vaccines while they are still hospitalised in neonatal units. There are no data regarding stool excretion of the RV1 rotavirus vaccine in premature babies - there is a theoretical risk of transmission of the vaccine virus to other babies in the unit (if there was inadequate staff hand washing). Some countries have therefore advised against immunisation of babies while in the neonatal unit. In the UK, however, the vaccine is being given in neonatal units, enabling evaluation of the vaccine in hospitalised premature babies.

This is an observational study of babies admitted to the neonatal unit at the John Radcliffe Hospital, Oxford University Hospitals NHS Trust who receive their first dose of rotavirus vaccine during their hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Participant's parent is willing and able to give informed consent for participation in the study.
* Current inpatient in the neonatal unit and expected to remain an inpatient for at least 14 days following immunisation with rotavirus vaccine.
* Due to receive rotavirus vaccination during their admission.
* Born at less than 37 completed weeks gestation (i.e. up to and including 36 weeks and 6 days)

Exclusion Criteria:

• Parent is listed on the study delegation log.

Ages: 8 Weeks to 15 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature babies receiving their first dose of rotavirus vaccine while an inpatient on the neonatal unit at the John Radcliffe Hospital, Oxford University Hospitals NHS Trust
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-12; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of days rotavirus vaccine can be detected in stool following immunisation | 24 months

SECONDARY OUTCOMES:
Measurement of serum and stool antibody to rotavirus vaccine following vaccination | 24 months
Number of adverse events following rotavirus vaccine | 12 months
Comparison of vaccine responses after categorisation based on GI microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pollard, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - Department of Paediatrics, University of Oxford, Oxford, Oxfordshire
  - Oxford University Hospitals NHS Trust, Oxford